CLINICAL TRIAL: NCT03196817
Title: Non-surgical Treatment of Carpal Tunnel Syndrome: Night Splint Versus Local Corticosteroid Infiltration: Clinical Randomized Trial
Brief Title: Non-surgical Treatment of Carpal Tunnel Syndrome: Night Splint Versus Local Corticosteroid Infiltration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Alvorada (Other)
Responsible Party: Principal Investigator, João Carlos Belloti, Clinical Professor, Hospital Alvorada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HAMJQ01
Record Dates: First submitted 2016-10-21; First posted 2017-06-23 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Random Allocation; Injections; Orthotic Devices
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — betamethasone-17,21-dipropionate; betamethasone sodium phosphate; Steroids

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carpal tunnel injection (Active Comparator): Carpal tunnel injection (infiltration) group of patients will be referred to the Hospital Alvorada to carry out steroid injection. The injection in carpal tunnel will be an association of 6.43 mg of betamethasone dipropionate, 2.63 mg of betamethasone disodium phosphate and 0.5 ml plus lidocaine 2%, totaling 1.5 ml.
  Interventions: Drug: betamethasone dipropionate, betamethasone disodium phosphate and lidocaine 2%
- Wrist splinting (Active Comparator): Wrist splinting will be use in the nigth time, remain the wrist in the 15th degree in extension, until its removal in the morning.
  Interventions: Device: Wrist splinting

INTERVENTIONS:
Drug: betamethasone dipropionate, betamethasone disodium phosphate and lidocaine 2% — 6.43 mg of betamethasone dipropionate, 2.63 mg of betamethasone disodium phosphate and 0.5 ml plus lidocaine 2%
  Other Names: Steroid injection
  Arms: Carpal tunnel injection
Device: Wrist splinting — Splinting only at night to maintain the wrist positioned in 15 degrees of extensionin.
  Other Names: wrist splints
  Arms: Wrist splinting

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common neuropathic compression syndrome of the upper limbs, caused by compression of the median nerve in the wrist. There is no gold standard for establishing the diagnosis of STC. The diagnosis can be based on clinical findings and electrodiagnostic tests. Treatment options can be divided into surgical and non-surgical procedures. Surgical interventions include open carpal tunnel release, mini incision or release of the endoscopic carpal tunnel. Nonsurgical include daily activities modification, oral anti-inflammatory drugs (NSAIDs), oral corticosteroids, splints, corticosteroid injections or other options (laser therapy, ultrasound or acupuncture)

The aim of this study is to compare randomly, conservative treatment for CTS with night splint of the wrist versus local infiltration of corticosteroids after a min-imum period of six months follow-up.

Patients will be divided into two groups: night orthesis group that will receive the prescription to purchase the orthesis and guide the use of it; and infiltration group of patients will be referred to the Moema Alvorada Hospital to carry out infiltration. These patients will be evaluated before application, one week, one month, three months and six months after intervention.

DETAILED DESCRIPTION:
This study will be developed in the service of medical residency of surgery and microsurgery of the hand of Alvorada hospital (São Paulo - SP).

The Study Design is Randomized clinical trial according to the CONSORT STATEMENT (http://www.consort-statement.org) standards.

The number of participants will initially be 84 patients.

Inclusion criteria:

Adult patients 40 years of age or older with four or more of the following clinical signs and symptoms suggested by Graham et al. (CTS-6):

1. Paresthesia in the territory of the median nerve.
2. Nocturnal paresthesia of the hand
3. Atrophy of the tenar musculature
4. Positive Tinel Signal
5. Positive Phalen Test
6. Loss of discrimination of 2 points

All patients will be diagnosed with electromyography (EMG). All participants will sign an Research Ethics Committee of this institution, after reading and explaining the study proposal.

Criteria for non-inclusion:

Previous treatment with corticosteroids and felling in the last 6 months Previous surgical treatment Associated traumatic or non-traumatic pathologies Hypersensitivity to corticosteroids. CTS secondary to another pathology. Refusal to Research Ethics Committe. Fixed paresthesia

Randomization and Allocation:

The allocation of patients to the infiltration or nocturnal orthosis groups will be performed using opaque and numbered envelopes on their outer face with consecutive numbers. The draw of the method, for each envelope, will be done randomly and sequentially, using randomization software (available at: http://www.random.org), after the randomization, the envelopes will be sealed. The sealed envelope, containing the patient's allocation group, will be opened only at the doctor's office after verification of the criteria for inclusion and signing of the Research Ethics Committee signature. The randomization procedure was performed by a person not directly involved in the study.

Sampe Size:

Considering the difference of 30% in the improvement of nocturnal paresthesia, 95% confidence interval and statistical power of 80%, we calculated a sample of 84 patients. At 6 months

Interventions

The patients included in this study will be attended at the Santa Cruz IV Ambulatory of hand surgery outpatient clinic. Patients with a diagnosis of CTS will be referred for evaluation in this outpatient clinic.

After confirmation of the diagnosis of CTS with the presence of four or more of the six criteria proposed by Graham and confirmation by the EMG and application of the inclusion and non inclusion criteria in the study, eligible patients will be informed about the nature and purpose of the study, by reading the Research Ethics Committee of this institution; after signing will be registered. Only after signing the Research Ethics Committee and the patient's registration will the opaque and sealed envelope containing the patient's allocation be opened. Patients in the nocturnal orthoses group will receive prescriptions for the purchase of the orthosis and guidance on use at the same moment of randomization. Patients in the infiltration group will be referred to the Hospital Alvorada de Moema to perform the infiltration at the same moment of randomization.

Infiltration technique:

Patient seated, with elbow resting on the table, supine wrist, relaxed in dorsiflexion, after asepsis and antisepsis care a needle will be inserted located on the ulnar border of the radial flexor tendon of the carpus, with an angle of 30º directed to the carpal tunnel , with an association of betamethasone dipropionate, betamethasone disodium phosphate {diprospan®}, plus lidocaine (xylocaina®).

Night immobilization:

During the night time, the patient will wear a forearm-palmar splint, where the wrist will remain in the 15th degree of extension, until its removal in the morning. The nocturnal orthosis should be used by study period .

Outcomes

Primary Outcomes:

1. Remission of nocturnal paresthesia after intervention - Evaluation to verify remission of nocturnal paresthesia, referred by the patient at the time of initial care.
2. Boston Questionnaire (Levine):

A questionnaire developed for the purpose of evaluating the severity of symptoms and the degree of manual ability of patients with CTS. This is a self-reported questionnaire that assesses the severity of symptoms and the functional status of patients.

Secondary Outcome Measures:

1. Visual Analogue Scale - EVA Pain Evaluation - The analogical visual scale of pain is formed by two bars, joined by a line with ten centimeters, that mark the beginning and the end. The start bar is "0" and indicates no pain. The end bar is the "10" and indicates the maximum pain. The patient was asked to register his pain with a stroke on that line joining the two bars. The gauging of the pain was performed by measuring the distance between the initial bar and the trait performed by the patient.
2. Graham Criteria - CTS-6 Assessment of improvement of graham's cervix, which are signs and symptoms used for the diagnosis of CTS

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 40 years or more,
* Have the diagnosis confirmed with electromyography (EMG),
* Four or more than six of the following clinical signs and symptoms suggested by Graham et al (CTS-6):

  * Paraesthesia in the territory of the median nerve.
  * Night hand paresthesia
  * Atrophy of thenar muscles
  * Positive Tinel Sign
  * Phalen Test Positive
  * Loss of two point discrimination
* Sign a Research Ethics Committe, after reading and explanation of the proposed study.

Non-inclusion criteria:

* Pretreatment with corticosteroids and splint
* Prior surgical treatment
* Traumatic or nontraumatic pathologies associated
* Hypersensitivity to corticosteroids
* CTS secondary to other pathology
* Refusal to sign a Research Ethics Committe.
* Fixed Paresthesia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Remission of symptoms | 6 months
  Remission of nocturnal paresthesia referred by the patient at six months the follow up.
Boston Questionnaire (Levine) | 6 months
  A questionnaire developed for the purpose of evaluating the severity of symptoms and the degree of manual ability of patients with CTS.

SECONDARY OUTCOMES:
Visual Analogue Scale - EVA Pain Evaluation | 6 months
  The analogical visual scale of pain is formed by two bars, joined by a line with ten centimeters, that mark the beginning and the end. The start bar is "0" and indicates no pain. The end bar is the "10" and indicates the maximum pain.
Graham Criteria - CTS-6 | 6 months
  Assessment of improvement of graham's cervix, which are signs and symptoms used for the diagnosis of CTS

CONTACTS AND LOCATIONS:
Overall Officials: Non-surgical T Infiltration, Principal Investigator — Hospital Alvorada
Locations (1):
- Jesus Queiroz junior, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chen PC, Chuang CH, Tu YK, Bai CH, Chen CF, Liaw M. A Bayesian network meta-analysis: Comparing the clinical effectiveness of local corticosteroid injections using different treatment strategies for carpal tunnel syndrome. BMC Musculoskelet Disord. 2015 Nov 19;16:363. doi: 10.1186/s12891-015-0815-8. PMID 26585378
- [Background] Ly-Pen D, Andreu JL, Millan I, de Blas G, Sanchez-Olaso A. Comparison of surgical decompression and local steroid injection in the treatment of carpal tunnel syndrome: 2-year clinical results from a randomized trial. Rheumatology (Oxford). 2012 Aug;51(8):1447-54. doi: 10.1093/rheumatology/kes053. Epub 2012 Mar 30. PMID 22467087
- [Background] Meems M, Den Oudsten B, Meems BJ, Pop V. Effectiveness of mechanical traction as a non-surgical treatment for carpal tunnel syndrome compared to care as usual: study protocol for a randomized controlled trial. Trials. 2014 May 22;15:180. doi: 10.1186/1745-6215-15-180. PMID 24886455
- [Background] Graham B, Regehr G, Naglie G, Wright JG. Development and validation of diagnostic criteria for carpal tunnel syndrome. J Hand Surg Am. 2006 Jul-Aug;31(6):919-24. PMID 16886290
- [Background] Peters-Veluthamaningal C, Winters JC, Groenier KH, Meyboom-de Jong B. Randomised controlled trial of local corticosteroid injections for carpal tunnel syndrome in general practice. BMC Fam Pract. 2010 Jul 29;11:54. doi: 10.1186/1471-2296-11-54. PMID 20670438
- [Background] Ucan H, Yagci I, Yilmaz L, Yagmurlu F, Keskin D, Bodur H. Comparison of splinting, splinting plus local steroid injection and open carpal tunnel release outcomes in idiopathic carpal tunnel syndrome. Rheumatol Int. 2006 Nov;27(1):45-51. doi: 10.1007/s00296-006-0163-y. Epub 2006 Jul 27. PMID 16871409
- [Background] Carlson H, Colbert A, Frydl J, Arnall E, Elliot M, Carlson N. Current options for nonsurgical management of carpal tunnel syndrome. Int J Clin Rheumtol. 2010 Feb;5(1):129-142. doi: 10.2217/IJR.09.63. PMID 20490348